CLINICAL TRIAL: NCT01226667
Title: Fixed Versus Flexible Dosing of Pregabalin in Patients With Fibromyalgia
Acronym: Flexdose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Osteoporosis Medical Center, Beverly Hills, CA (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SLS2009001
Record Dates: First submitted 2010-10-01; First posted 2010-10-22 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; lyrica; pregabalin
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flexible Dose (Active Comparator): flexibly dosed pregabalin given BID (75-300 mg/d) increased gradually over 4 weeks then maintained at that same dosing for 4 weeks
  Interventions: Drug: Pregabalin
- Fixed Dosing (Active Comparator): 75 mg BID for one week and increased to 150 mg BID for 7 weeks
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Fixed dosing of pregabalin: Week 1: 75 mg bid. Weeks 2 - 8: 150 mg bid. Week 9 (Days 57-60 and Days 61-63): 75 mg bid.
  Flexible dosing of pregabalin: Week 1: placebo in the AM and 75 mg nightly; Week 2: placebo in the AM and 150 mg nightly.; Week 3 placebo in the a.m., 225 mg nightly; Weeks 4 - 8 placebo in the a.m., 300 mg nightly. Week 9 (Days 57-60) placebo in the a.m,, 150 mg bid nightly and Days 61-63: placebo in the a.m., and 75 mg bid nightly.

SUMMARY:
A 9-week randomized double-blind, multi-center study of 172 patients, who after 1 week baseline evaluation are randomized to either fixed dose pregabalin starting at 75 mg BID for one week and increased to 150 mg BID for 7 weeks or flexibly dosed pregabalin given BID (75-300 mg/d) increased gradually over 4 weeks then maintained at that same dosing for 4 weeks.It is proposed that use of flexible dosing combined with nightly dosing would have similar pain relief to fixed dosing, would improve adherence, would have less side effects and would be more likely to improve sleep.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of fibromyalgia by ACR criteria
* ambulatory patients
* complete of 5 pain diaries during 1 week evaluation
* other inclusion criteria may apply

Exclusion Criteria:

* pregnant or of childbearing potential not using contraceptives
* use of pregabalin in the past
* concomitant use of opioids or gabapentin
* estimated creatinine clearance less than 60
* other criteria may apply

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Pain score evaluation by NRS | 8 weeks
  Least square mean change in Fibromyalgia pain at 8weeks compared to baseline utilizing an 11 point numerical rating scale daily pain diary (0 = no pain to 10 =worst possible pain) performed at daily awakening.

SECONDARY OUTCOMES:
Patient Global Impression of Change | At weeks 4 and 8
Discontinuation rate | 9 weeks
  Discontinuation rates due to lack of efficacy and discontinuation rates due to adverse event.
Improvements in Wolfe Symptom Severity Score | 9 weeks
  Wolfe Symptom Severity scales for pain, fatigue, trouble sleeping, trouble with anxiety or depression, trouble thinking or remembering, overall FM severity, problems awaking feeling unrefreshed

CONTACTS AND LOCATIONS:
Overall Officials: Keaton Nasser, Study Director — Osteoporosis Medical Center; Stuart L Silverman, M.D., Principal Investigator — Osteoporosis Medical Center
Locations (5):
- United States (5):
  - David Silver MD Inc, Beverly Hills, California
  - Stuart L Silverman MD Inc., Beverly Hills, California
  - Talbert Medical Group, Huntington Beach, California
  - Catalina Pointe Clinial Research, Tucson, California
  - Affilaites in Medical Specialty, West Hills, California

REFERENCES:
- [Derived] Nasser K, Kivitz AJ, Maricic MJ, Silver DS, Silverman SL. Twice daily versus once nightly dosing of pregabalin for fibromyalgia: a double-blind randomized clinical trial of efficacy and safety. Arthritis Care Res (Hoboken). 2014 Feb;66(2):293-300. doi: 10.1002/acr.22111. PMID 23983064